CLINICAL TRIAL: NCT02806011
Title: Long-term Follow-up Study of Livercellgram in Alcoholic Liver Cirrhosis Patients Who Completed Livercellgram Phase 2 Study
Brief Title: Long-term Follow-up Study of Livercellgram in Alcoholic LC Patients Who Completed Livercellgram Phase 2 Study
Status: Completed | Type: Observational
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PMC-P-002-01
Record Dates: First submitted 2016-06-15; First posted 2016-06-20 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Alcoholic Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- no Intervention: Long-term follow up of no intervention group
- 1-time injection group: Long-term follow up of 1-time injection group
- 2-time injection group: Long-term follow up of 2-time injection group

SUMMARY:
This is a 5-year (+30 days) long term follow up study to evaluate the safety of Livercellgram in subject who participated in and completed the Livercellgram Phase 2 trials (refer to ClinicalTrials.gov.Identifier: NCT01875081).

DETAILED DESCRIPTION:
This is a 5-year (+30 days) long term follow up study to evaluate the safety of Livercellgram in subject who participated in and completed the Livercellgram Phase 2 trials (refer to ClinicalTrials.gov.Identifier: NCT01875081).

This trial is planned to evaluate the safety of Livercellgram in patients with alcoholic liver cirrhosis. Subjects who signed this follow-up observation informed consent form will participate in a safety assessment (tumor marker test, occurrence of adverse events and serious adverse events, clinical laboratory tests, vital sign, physical examinations.).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who treated with Livercellgram and completed the Livercellgram phase 2 study.
2. Subjects who can agree to participate in the long term observation study by oneself.

Exclusion Criteria:

* Not Applicable

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have completed the Livercellgram phase 2 study and can agree to participate in the long term observation study by oneself.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2016-05; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Safety Evaluation assessed by Tumor Marker Test, Adverse Events and Serious Adverse Events, Clinical Laboratory Tests, Vital Signs, and Physical Examinations | 5-year(+30 days)
  1. Tumor Marker Test
  2. Occurrence of Adverse Events and Serious Adverse Events
  3. Clinical Laboratory Tests
  4. Vital Sign
  5. Physical Examinations

CONTACTS AND LOCATIONS:
Overall Officials: Soon Koo Baik, M.D.,Ph.D, Principal Investigator — Wonju Severance Christian Hospital
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, South Korea